CLINICAL TRIAL: NCT03808857
Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of GB226 in Treatment of Recurrent or Metastatic Cervical Cancer Patients With PD-L1 Positive Who Failed in Platinum-based Chemotherapy
Brief Title: A Study in Recurrent or Metastatic Cervical Cancer Patients With PD-L1 Positive
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-008
Record Dates: First submitted 2018-12-27; First posted 2019-01-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer
Keywords: recurrent Metastatic Cervical Cancer; platinum
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226 (Experimental): Geptanolimab Injection,3mg/kg once per 2 weeks
  Interventions: Biological: GB226

INTERVENTIONS:
Biological: GB226 — GB226 is administrated at the dose of 3mg/kg, once per 2 weeks (±3 days), and distributed in 100ml of 0.9% sodium chloride solution. The concentration of GB226 shall be strictly controlled at 1mg/ml~10mg/ml, the duration is 60 min (±10 min) for the first infusion of the drug, and can be reduced to 30 min (±10 min) for the subsequent infusion of the drug if there is infusion related adverse reaction.
  Other Names: Geptanolimab

SUMMARY:
This study is a multi-center, prospective, open-label, single-arm phase II clinical study to evaluate the efficacy, safety and immunogenicity of GB226 in treatment of recurrent or metastatic cervical cancer patients with PD-L1 positive who failed in platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old;
* 2. Understand the steps and contents of the study, and voluntary to sign the written informed consent form;
* 3. Recurrent or metastatic cervical cancer diagnosed by histology or cytology;
* 4. Recurrent or metastatic after receiving at least first-line platinum base chemotherapy (≥1 period) (Subjects who progress or recur during or within 6 months after the end of platinum-based new adjuvant or adjuvant chemotherapy are deemed to have received first-line treatment);
* 5. Subjects must have at least one measurable target lesion (lesion with longest diameter ≥10mm, or lymph node with short diameter ≥15mm) tested by CT or MRI according to the RECIST 1.1 criteria;
* 6. Expected survival period ≥3 months;
* 7. ECOG score 0-1 point;
* 8. Subjects shall provide sufficient formalin fixed paraffin embedded (FFPE) specimens or sections prepared from tumor archived tissues or fresh tissues that meet the test criteria, and are willing to perform biopsy of tumor tissues for test of PD-L1 if needed. The archived tissue shall be a representative tumor specimen within three years, or unstained serial sections (not less than 4) of the newly cut FFPE tumor tissue within six months, and the above-mentioned specimens related pathology reports shall also be provided. Fresh tissue specimens can be obtained by resection, core needle biopsy, excision, stamping or forceps biopsy (more than 100 tumor cells must be guaranteed); samples are not accepted for fine needle puncture and liquid based cytology test (TCT) (namely, the samples lack of complete tissue structure thus to only provide cell suspension and/or cell smear); decalcified bone metastatic tumor samples are not accepted. For core-needle biopsy specimens, at least 3 single paraffin embedded specimens shall be submitted for evaluation. For patients with PD-L1 negative in initially archived tumor tissue samples, biopsy can be performed during screening with the patients' consent to provide fresh tissue prepared paraffin blocks or sections for retest of PD-L1 status, and the qualification of this study is met if any kind of tumor tissue samples have positive results;
* 9. The values of laboratory tests performed during screening shall meet the following criteria:

  * Blood routine test (No blood transfusion within 14 days before test, no use of G-CSF, no use of drug correction);

    1. Hemoglobin (HGB) ≥90 g/L;
    2. Absolute neutrophil count (ANC) ≥1.5×109/L;
    3. Blood platelet (PLT) ≥100×109/L；
  * Biochemical test

    1. Total bilirubin (TBIL) ≤1.5× Upper limit of normal (ULN) (Gilbert syndrome allowance ≤5×ULN);
    2. Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (if liver metastasis exists, ALT and AST ≤5×ULN);
    3. Serum creatinine (Cr) ≤1.5×ULN or endogenous creatinine clearance rate ≥50mL/min (Cockcroft-Gault formula);
* 10. Thyroid function index: Thyroid-stimulating hormone (TSH) and free thyroxine (FT3/FT4) are in normal range; Subjects could be enrolled if FT3/FT4 in the normal range,and TSH without the normal range;
* 11. Women who are not pregnant within 7 days before administration of study drug; women in child-bearing period shall agree to use medically approved effective contraception throughout the whole study period and within 6 months after completion of study;
* 12. Subjects can be followed up on schedule, able to communicate well with the investigator, and able to complete the study in accordance with the requirements of this study.

Exclusion Criteria:

* 1. Patient with other previous malignancies (except the cured skin basal cell carcinoma or squamous cell carcinoma) shall not participate in this study unless she experiences a "complete response" for at least 5 years before enrollment, and it is estimated that no other anti-tumor therapy will be required during the whole study;
* 2. Active central nervous system (CNS) metastasis, including symptomatic brain metastasis or meningeal metastasis or spinal cord compression, etc.; asymptomatic brain metastasis can be enrolled (no progression within at least 4 weeks after radiotherapy and/or no postoperative neurological symptoms or signs, no need for treatment with glucocorticoid, anticonvulsant drugs or mannitol);
* 3. Experienced systemic chemotherapy, radial/extensive radiotherapy, targeted therapy, anti-tumor biotherapy (e.g. tumor vaccine, cytokine or growth factor, etc.) within 28 days before administration of study drug, or experienced local palliative radiotherapy within 14 days;
* 4. Less than 14 days before the study was conducted with major surgery or severe trauma(Subjects could be enrolled ,except for skin or percutaneous biopsy with local anesthesia ,and recovered within 7 days);
* 5. Received corticosteroids (prednisone > 10 mg/day or equivalent dose) or other immunosuppressive drugs within 14 days before administration of study drug;
* 6. Have active, known history of autoimmune disease, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc. other than type I diabetes mellitus, hypothyroidism controlled only by hormone replacement therapy, skin diseases (e.g. vitiligo) requiring no systemic treatment and controlled celiac disease;
* 7. Complications requiring the treatment with immunosuppressive drugs, or complications requiring systemic treatment at the dose with immunosuppressive effects (prednisone > 10mg/day or equivalent dose to similar drug); in the absence of active autoimmune disease, inhaling or local administration of steroids and prednisone at dose > 10mg/day or equivalent dose to similar drug are allowed;
* 8. Uncontrolled hypertension (systolic pressure >140 mmHg and/or diastolic pressure > 90 mmHg) or pulmonary hypertension or unstable angina pectoris; underwent myocardial infarction, bypass or stent surgery within 6 months before administration; have a history of grade 3-4 chronic heart failure that meets the criteria of New York Heart Association (NYHA); Valvular heart disease with clinical significance; severe arrhythmia requiring treatment, including QTc interval ≥ 470 ms (calculate by Fridericia formula); left ventricular ejection fraction (LVEF) < 50%; Cerebral vascular accident (CVA) or transient ischemic attach (TIA) within 6 months before administration, etc.;
* 9. Complicated with other serious medical disease, including but not limited to uncontrolled diabetes mellitus, active gastrointestinal ulcers, active hemorrhage, etc.;
* 10. Subjects suffering from active infections that require systemic treatment;
* 11. Patients with previous or present infection with active tuberculosis;
* 12. Have the previous history of interstitial pulmonary disease;
* 13. Uncontrollable symptomatic dropsy of serous cavity, such as ascites, pleural effusion or pericardial effusion;
* 14. Human immunodeficiency virus antibody (HIV-Ab) and Treponema pallidum positive; hepatitis C antibody (HCV-Ab) positive, and hepatitis C virus RNA quantification > the upper limit of normal of test unit; hepatitis B surface antigen (HBsAg) positive, and hepatitis B virus test value > the upper limit of normal of test unit;
* 15. Adverse events caused by previous treatment have not recovered to grade 1 or below (CTCAE5.0) (except the grade 2 neurotoxicity caused by alopecia and chemotherapeutics);
* 16. Have been treated with anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4 antibody (or any other antibodies acting on T cell co-stimulation or checkpoint pathway);
* 17. Used live vaccine or attenuated vaccine within 28 days before administration of study drug;
* 18. Used other study drugs or study devices within 30 days before administration of study drug;
* 19. Patients with a history of drug addiction or drug abuse upon inquiry;
* 20. Patients with previous definite neurological or mental disorders, such as epilepsy, dementia, poor compliance;
* 21.Lactating women who do not agree to stop breastfeeding ;
* 22. Known allergy to recombinant human PD-1 monoclonal antibody or any of its excipients; known history of allergic disease or severe allergic constitution;
* 23. Patients who are not suitable for participating in this study due to other various reasons upon investigator's opinions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 2 years
  To evaluate the efficacy of GB226 as defined by objective response rate, in patients with recurrent or metastatic cervical cancer.

SECONDARY OUTCOMES:
Disease control rate,DCR | 2 years
  To evaluate the efficacy of GB226 as defined by overall response rate, in patients with recurrent or metastatic cervical cancer.
Time to response, TTR | 2 years
  To evaluate the efficacy of GB226 as defined by time to response in patients with recurrent or metastatic cervical cancer.
Duration of response, DOR | 2 years
  To evaluate the duration of response (DOR) of GB242 in patients with recurrent or metastatic cervical cancer.
Progression-free survival, PFS | 2 years
  To evaluate the efficacy of GB226 as defined by progression-free survival, in patients with recurrent or metastatic cervical cancer.
Overall survival, OS | 2 years
  To evaluate the duration from the first administration to death because of any reason in patients with recurrent or metastatic cervical cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China